CLINICAL TRIAL: NCT01417468
Title: Instructional Design Strategies to Support Adult Patients/Students (Civilian & Military) With Traumatic Brain Injury (TBI).
Brief Title: How Well do Patients With Traumatic Brain Injury Learn New Material Using Learning Styles in Online Science Classrooms?
Acronym: CVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Vision Development, New Market, Maryland (Other)
Responsible Party: Principal Investigator, Mark Pettinato, Principal Investigator, Center for Vision Development, New Market, Maryland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CVDMaryland-001
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Brain Injuries; Brain Injuries, Traumatic; Injury, Brain, Traumatic; Traumatic Brain Injury; Brain Injury, Chronic
Keywords: Cognitive Rehabilitation; Learning Styles; Learning Modes; Learning Modalities; Multiple Intelligences; Educational Intervention; Instructional Design
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Brain Injury, Chronic | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLSI - Known (Experimental): Participants will be assigned to a specific learning group via the Canfield Learning Style Inventory (CLSI).
  Interventions: Behavioral: CLSI, MI, CR
- CLSI - Unknown (Active Comparator): Participants will be assigned to a traditional learning group (Control).
  Interventions: Behavioral: CLSI - Unknown

INTERVENTIONS:
Behavioral: CLSI, MI, CR — (CLSI) Canfield Learning Styles Inventory (MI) Multiple Intelligences (CR) Cognitive Rehabilitation
  Other Names: Canfield Learning Styles Inventory; Multiple Intelligences; Cognitive Rehabilitation
  Arms: CLSI - Known
Behavioral: CLSI - Unknown — (CLSI) Canfield Learning Styles Inventory (MI) Multiple Intelligences (CR) Cognitive Rehabilitation
  Other Names: Canfield Learning Styles Inventory; Multiple Intelligences; Cognitive Rehabilitation
  Arms: CLSI - Unknown

SUMMARY:
The purpose of this study is to determine whether learning styles are effective in the treatment of traumatic brain injury (TBI) in an educational environment.

DETAILED DESCRIPTION:
The purpose of this study is to determine the learning outcome and effectiveness of instructional design strategy using Canfield's learning styles and Gardner's Multiple Intelligences to accommodate TBI-induced cognitive impairments in an online science learning environment.

ELIGIBILITY:
Inclusion Criteria:

1. People who have been diagnosed with Mild Traumatic Brain Injury (TBI).
2. People who are able to understand and sign an informed consent form.
3. People who have no other known neurological disorder (e.g. aphasia, stroke).
4. All participants must be 18-50 years old.
5. Be able to speak and understand English, and
6. Have use of a computer (Mac or Windows) and internet (www) access.

Exclusion Criteria:

1. Don't meet the inclusion Criteria
2. Other known neurological disorder (e.g. aphasia, stroke).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-02 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Learning Effectiveness | 3 Months
  This study will explore the use of a cognitive rehabilitation approach as suggested by Gardner's Multiple Intelligences for its potential application to online course design for brain injured patients/students. It involves designing instruction for a science unit based on four of Canfield's learning styles.

CONTACTS AND LOCATIONS:
Overall Officials: Mark C. Pettinato, M.S., Principal Investigator — Capella University
Locations (1):
- Center for Vision Development - (Research is being conducted online), New Market, Maryland, United States

REFERENCES:
- [Background] Canfield, A. (1980). Learning styles inventory manual. Ann Arbor, MI: Humanics Media. Pashler, H.; McDaniel, M.; Rohrer, D.; Bjork, R. (2009).